CLINICAL TRIAL: NCT05358210
Title: The Clinical and Physiological Effects of Blueberry Consumption in Older Adults
Brief Title: Effects of Blueberries in Older Adults
Acronym: BnD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: U.S. Highbush Blueberry Council (Other)
Responsible Party: Principal Investigator, Kenneth Mukamal, Associate Section Chief for Research, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021P001034
Record Dates: First submitted 2022-04-21; First posted 2022-05-03 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Blood Pressure; Orthostatic Hypotension; Vascular Diseases
Keywords: Blueberries; Dates; Older Adults; Blood pressure; Fruit; Vascular health; Dietitian
MeSH Terms: conditions — Hypotension, Orthostatic; Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Individual, parallel-design, randomized trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blueberry Consumption (Experimental): Randomized participants will consume 1 cup of frozen blueberries, provided by the trial, daily for 12 weeks.
  Interventions: Behavioral: Blueberry Consumption
- Dried Date Consumption (Active Comparator): Randomized participants will consume 2-3 dried dates, provided by the trial, daily for 12 weeks.
  Interventions: Behavioral: Dried Date Consumption

INTERVENTIONS:
Behavioral: Blueberry Consumption — Participants will consume 1 cup of frozen blueberries daily for the 12 weeks of the intervention. The study dietitian will provide educational materials and monitor compliance through weekly check-ins. Participants will be instructed to avoid all other high-anthocyanin foods including other berries, cherries, currants, cabbage, red wine, and eggplant.
  Arms: Blueberry Consumption
Behavioral: Dried Date Consumption — Participants will consume 2-3 dried dates daily for the 12 weeks of the intervention, an isocaloric portion of fruit compared to the blueberry group. The study dietitian will provide educational materials and monitor compliance through weekly check-ins. Participants will be instructed to avoid all other high-anthocyanin foods including blueberries, other berries, cherries, currants, cabbage, red wine, and eggplant.
  Arms: Dried Date Consumption

SUMMARY:
This randomized, parallel-design trial will evaluate specific clinical and physiological effects of whole blueberries in adults 70 years of age or older.

DETAILED DESCRIPTION:
Although much is already known about the benefits of a healthy diet for the prevention of a wide range of chronic diseases, including the particular health benefits of anthocyanin-rich foods, these effects have been examined with much less frequency in older adults, who tend to be excluded from formal feeding studies and, until recently, have represented a small proportion of ongoing cohort studies. The proposed study will randomize approximately 46 women and 24 men, representative of the proportion of elderly women and men in the U.S. to consume either:

1. 1 cup of frozen blueberries daily for 12 weeks

   or
2. 2-3 dried dates daily for 12 weeks.

Dates were chosen as a control food because they contain negligible polyphenols, proportionately high caloric content, and a convenient form for storage. After the 12-week intervention, researchers will repeat in-person study assessments from baseline.

ELIGIBILITY:
Inclusion Criteria:

* 70 years old
* Independent-living

Exclusion Criteria:

* Cardiovascular event or procedure within 3 months of randomization
* AHA Class III-IV heart failure
* Intolerance or allergy to blueberries or dates
* History of gastric bypass surgery
* Any planned hospitalization or vacation in the ensuing 4 months
* Any current cancer treatment
* End-stage renal disease
* Any organ transplant
* Uncontrolled diabetes mellitus with hemoglobin A1c >9%
* Systolic blood pressure >200 mmHg
* Inability to provide personal informed consent (e.g. cognitive impairment)
* Investigator concern

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure Monitoring | 12 weeks after randomization
  24-hour wake-time ambulatory blood pressure monitoring
Orthostatic Hypotension | 12-weeks after randomization
  Supine and standing blood pressure
Lower Extremity Functioning | 12 weeks after randomization
  Short Physical Performance Battery
Cognition | 12 weeks after randomization
  Cogstate Brief Battery of four core cognitive domains: processing speed, attention, visual learning, and working memory

SECONDARY OUTCOMES:
Number of Self-Reported Falls | Weekly for 12 weeks between baseline and follow-up
  Investigators will administer the Fall Follow-Up Questionnaire from the Study to Understand Fall Reduction and Vitamin D in You (STURDY) to participants that self-report falls to record details on each fall.
Grip Strength | 12 weeks after randomization
  Bilateral grip strength measured by a dynamometer
Sleep | 12 weeks after randomization
  Pittsburgh Sleep Quality Index. The 19 self-rated items are combined to form 7 "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The 7 component scores are then added to yield one "global score", with a range of 0-21 points, "0" indicating no difficulty and "21" indicated severe difficulties in all sleep areas.
Incontinence | 12 weeks after randomization
  Questionnaire for Urinary Incontinence Diagnosis. The first 3 items focus on stress incontinence symptoms and the last 3 on urge incontinence symptoms. Each item includes 6 frequency-based response options, which are scored from 0 to 5 points. Scores are calculated in an additive fashion, resulting in separate Stress and Urge score, each ranging from 0-15 points. Higher scores indicate more severe incontinence symptoms.
Cardiac Ectopy | 12 weeks after randomization
  Number of participants with atrial premature beats detected by a 24-hour Holter monitor
Troponin T (HS) | 12 weeks after randomization
  Measured in blood sample
High Density Lipoprotein Cholesterol | 12 weeks after randomization
  Measured in fasted blood as part of a lipid panel
Total Cholesterol | 12 weeks after randomization
  Measured in fasted blood as part of a lipid panel
Derived Low Density Lipoprotein Cholesterol | 12 weeks after randomization
  Measured in fasted blood as part of a lipid panel
Triglycerides | 12 weeks after randomization
  Measured in fasted blood as part of a lipid panel
Estimated Glomerular Filtration Rate (eGFR) | 12 weeks after randomization
  Measured in blood as part of basic metabolic panel
Albumin-to-Creatinine Ratio | 12 weeks after randomization
  Measured in a spot urine sample to detect albuminuria
Fructosamine | 12 weeks after randomization
  Measured in blood to estimate glucose levels over the previous 2-3 weeks.
Free Fatty Acids | 12 weeks after randomization
  Measured in blood samples
C-Reactive Protein (CRP) | 12 weeks after randomization
  Measured concentration in blood in response to inflammation
C-terminal telopeptide of type 1 collagen | 12 weeks after randomization
  Measured in blood samples to assess bone turnover
T-Cell Receptor Portfolio | 12 weeks after randomization
  Adaptive Immune Receptor Repertoire sequences in blood samples
Immune System Diversity | 12 weeks after randomization
  Measure in blood samples to show diversity of immune sequences

OTHER OUTCOMES:
Liver Enzymes | 12 weeks after randomization
  Measuring AST and ALT in blood samples
Total and Direct Bilirubin | 12 weeks after randomization
  Measured in blood samples
Fasting Glucose | 12 weeks after randomization
  Measured in blood samples
Fasting Insulin | 12 weeks after randomization
  Measured in blood samples
White Blood Cell Count | 12 weeks after randomization
  Measured in blood samples as part of complete blood count

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Mukamal, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Center Communities of Brookline (CCB), Brookline, Massachusetts
  - NewBridge on the Charles, Dedham, Massachusetts

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT05358210/Prot_000.pdf